CLINICAL TRIAL: NCT06479343
Title: Efficacy and Safety of the Liquid Embolic System (Tonbridge) for Endovascular Treatment of Cerebrovascular Malformations: a Prospective, Multi-center, Randomized, Parallel Positive Controlled, Non-inferiority Trial
Brief Title: Efficacy and Safety of the Liquid Embolic System (Tonbridge) for Endovascular Treatment of Cerebrovascular Malformations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZTQ202401
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Arteriovenous Malformations
MeSH Terms: conditions — Intracranial Arteriovenous Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liquid Embolic System (Tonbridge) (Experimental)
  Interventions: Device: Liquid Embolic System (Tonbridge)
- Onyx Liquid Embolic System (Medtronic) (Active Comparator)
  Interventions: Device: Onyx Liquid Embolic System (Medtronic)

INTERVENTIONS:
Device: Liquid Embolic System (Tonbridge) — Endovascular treatment with Liquid Embolic System (Tonbridge).
  Arms: Liquid Embolic System (Tonbridge)
Device: Onyx Liquid Embolic System (Medtronic) — Endovascular treatment with Onyx Liquid Embolic System (Medtronic).
  Arms: Onyx Liquid Embolic System (Medtronic)

SUMMARY:
The purpose of this study is to verify the efficacy and safety of the Liquid Embolic System (Tonbridge Medical Tech. Co., Ltd. (Suzhou)) for the treatment of cerebrovascular malformations.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized, parallel positive controlled, non-inferiority trial. This clinical trial is conducted at more than 2 centers in China, and patients who intend to be treated with liquid embolic system for cerebrovascular malformations are enrolled. Eligible patients are randomized into experimental group using Liquid Embolic System (Tonbridge) or control group using Onyx Liquid Embolic System (Medtronic) in a 1:1 ratio. The purpose of this study is to evaluate the effectiveness and safety of the Liquid Embolic System (Tonbridge).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years, any gender;
* Subject is suitable for endovascular treatment of cerebrovascular malformations;
* Subject is able to understand the purpose of the study, shows sufficient compliance with the study protocol and provides a signed informed consent form.

Exclusion Criteria:

* Intracranial hemorrhage within 1 month prior to treatment;
* The targeted embolization area needs to receive other treatments (surgical resection, SRS, other embolic materials) at the same time;
* Combination of other cerebrovascular malformations, such as cavernous vascular malformation;
* Severe stenosis or occlusion of cerebral feeding artery requiring surgical intervention;
* Intracranial tumor requiring surgical intervention;
* mRS score≥3;
* Heart, lung, liver and renal failure or other severe diseases;
* Known bleeding tendency, such as coagulation dysfunction (INR>1.5);
* Known allergy to DMSO and contrast media, or contraindication to anticoagulant therapy;
* Pregnant or breastfeeding women, or who plan to become pregnant during the study;
* Subject is participating in other drug or medical device clinical trials at the time of signing informed consent;
* Other conditions judged by the investigators as unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Targeted Embolization Satisfaction Rate | intra-procedure
  Targeted embolization satisfaction is defined as achieving ≥50% occlusion of the targeted embolized area after treatment with liquid embolic system, which is determined by immediate postoperative cerebrovascular DSA.

SECONDARY OUTCOMES:
mRS score | 1 month±7 days, 3 months±30 days, 6 months±30 days, 12 months±45 days post-procedure
  mRS scores are assessed at each evaluation time point.
GOS score | 1 month±7 days, 3 months±30 days, 6 months±30 days, 12 months±45 days post-procedure
  GOS scores are assessed at each evaluation time point.
Operation satisfaction rate | intra-procedure
  The 5-point Likert scale is used to evaluate operation satisfaction from three aspects: visualization, diffusion, and microcatheter withdrawal. "Operation satisfaction rate" is defined as the proportion of investigational devices or comparators with Likert score≥12 points.
Incidence of major adverse events (MAEs) | 1 month±7 days, 3 months±30 days post-procedure
  MAEs are defined as intracranial hemorrhage and ischemic complications. Intracranial hemorrhage included intraoperative hemorrhage (puncture of blood-supplying arteries by catheters or guidewires, rupture of nidus, and injury to blood vessels during withdrawal of catheters) and delayed symptomatic hemorrhage in the postoperative period; and ischemic complications included intraoperative ischemic complications (displacement of liquid embolic agents, thrombosis, and so on) and postoperative symptomatic ischemic stroke. "Incidence of major adverse events" is the proportion of subjects with adverse events using the investigational device or the comparator.
Incidence of adverse events (AEs) | 1 month±7 days, 3 months±30 days, 6 months±30 days, 12 months±45 days post-procedure
  "Incidence of adverse events" is the proportion of subjects with adverse events using the investigational device or the comparator.
Incidence of serious adverse events (SAEs) | 1 month±7 days, 3 months±30 days, 6 months±30 days, 12 months±45 days post-procedure
  "Incidence of serious adverse events" is the proportion of subjects with serious adverse events using the investigational device or the comparator.
Incidence of device deficiency | 3 months±30 days, 6 months±30 days, 12 months±45 days post-procedure
  Device deficiency is the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems and malfunctions.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Zhang, Principal Investigator — Xuanwu Hospital, Beijing
Locations (14):
- China (14):
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Xuanwu hospital Capital Medical University, Beijing
  - Sichuan Academy of Medical Sciences Sichuan Provincial People's Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Anhui Provincial Hospital, Hefei
  - Jining No.1 People's Hospital, Jining
  - Tongji Hospital Tongji Medical College of HUST, Wuhan

IPD SHARING:
Plan to Share IPD: No